CLINICAL TRIAL: NCT02051062
Title: Pharmacokinetics of Botulism Antitoxin Heptavalent (A, B, C, D, E, F, G) - (Equine) (BAT®) in Pediatric Patients With a Confirmed or Suspected Exposure to Botulinum Neurotoxin
Brief Title: BT-011 Pharmacokinetics of Botulism Antitoxin Heptavalent in Pediatric Patients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BT-011
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Botulism
Keywords: Pharmacokinetics; BAT; Pediatric
MeSH Terms: conditions — Botulism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Blood sample collection (Experimental): One to three 5 mL blood samples will be collected from pediatric participants treated with BAT product ideally 6-24 hours after administration, but within a maximum of 32 hours after administration.
  Interventions: Biological: Blood sample collection

INTERVENTIONS:
Biological: Blood sample collection — One to three 5 mL blood samples will be collected from pediatric participants treated with BAT product ideally 6-24 hours after administration but within a maximum of 32 hours after administration.

SUMMARY:
The purpose of this study is to verify the pediatric dosing recommendations for BAT product in pediatric patients that are treated with BAT product due to a confirmed or suspected case of botulism. A minimum of one serum sample should be collected but whenever feasible additional serum samples (up to three per enrolled participant) may be collected from the participant or obtained from surplus standard of care samples, if available, within 32 hours after BAT product administration. Safety of the BAT product will also be evaluated. Emergent will follow-up with the physician by telephone after 30 days post-BAT product administration to collect AEs, SAEs, and unanticipated events.

DETAILED DESCRIPTION:
Primary Objective: To collect blood from pediatric participants to analyze the pharmacokinetics (PK) of BAT product to verify the current US FDA-approved pediatric dosing recommendations for BAT product.

Safety Objective: To evaluate the safety of BAT product in pediatric participants.

Protocol Design: This is a single arm, multi-site PK study in pediatric patients treated with BAT product.

Pharmacokinetic Parameters: The serum concentrations of BAT product obtained will be modeled using a population PK approach based on a previously developed model for BAT serotypes A through G in healthy adult human participants.

Safety Endpoints: The incidence of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESI) that occur within 30 days after BAT product administration. In this study hypersensitivity/allergic reactions including serum sickness, febrile reactions, and hemodynamic instability and bradycardia, as well as reports of an infectious disease transmission will be included as AESI.

ELIGIBILITY:
Inclusion Criteria:

1. Legally authorized representative is able and willing to voluntarily provide informed consent and patients to provide assent, if applicable.
2. Pediatric participants (age groups: birth to <two years, two to <six years, and six to <12 years).
3. Treatment with BAT product (initial dose only).
4. Blood sample can be collected (or standard of care sample scavenged) within 32 hours of completion of BAT product infusion.

Exclusion Criteria:

1. If the 5 mL blood sample volume is deemed, at the discretion of the investigator, to be unsafe based on patient weight or condition of health.
2. History of treatment with BabyBIG or other botulism antitoxin within the past 90 days.

Ages: 1 Day to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Margin of PK Equivalence for 90% Survival | ideally up to 32 hours post-BAT product administration
  Margin of PK equivalence (MOE) for 90% survival relative to the healthy adult PK model, calculated to verify the appropriateness of administered pediatric dose. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.

SECONDARY OUTCOMES:
Area Under Concentration Curve From Time 0 to Last Measurable Concentration [AUC0-t] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameter: Estimated area under the serum concentration-time curve from time 0 to the last measurable serotype A concentration [AUC0-t]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Area Under Concentration Curve From Time 0 to Infinity [AUC0-inf] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameter: Estimated area under the serum concentration-time curve from time 0 to infinity [AUC0-inf]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Between Subject Variability [BSV] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameter: Between subject variability [BSV]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Maximum Serum Serotype A Concentration [Cmax] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameters: Estimated maximum serum serotype A concentration [Cmax]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Systemic Clearance [CL] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameters: Estimated systemic clearance [CL]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Intercompartmental Clearance [CLd] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameters: Estimated intercompartmental clearance [CLd]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Central Volume of Distribution [Vc] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameters: Estimated central volume of distribution [Vc]. All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.
Peripheral Volume of Distribution [Vp] | ideally up to 32 hours post-BAT product administration
  Pharmacokinetic Parameters: Estimated peripheral volume of distribution [Vp]). All collected samples of sufficient volume will be used provided both the BAT dosing time and sample collection time are known, even if outside the 32 hour collection window.

OTHER OUTCOMES:
Safety: AEs | Day 1 to Day 30
  Number of AEs that occur within 30 days after BAT product administration
Safety: SAEs | Day 1 to Day 30
  Number of SAEs that occur within 30 days after BAT product administration
Safety: AESI | Day 1 to Day 30
  Number of AESI that occur within 30 days after BAT product administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Representative, Study Director — Emergent BioSolutions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Richardson JS, Parrera GS, Astacio H, Sahota H, Anderson DM, Hall C, Babinchak T. Safety and Clinical Outcomes of an Equine-derived Heptavalent Botulinum Antitoxin Treatment for Confirmed or Suspected Botulism in the United States. Clin Infect Dis. 2020 Apr 15;70(9):1950-1957. doi: 10.1093/cid/ciz515. PMID 31209461
- [Background] Parrera GS, Astacio H, Tunga P, Anderson DM, Hall CL, Richardson JS. Use of Botulism Antitoxin Heptavalent (A, B, C, D, E, F, G)-(Equine) (BAT(R)) in Clinical Study Subjects and Patients: A 15-Year Systematic Safety Review. Toxins (Basel). 2021 Dec 27;14(1):19. doi: 10.3390/toxins14010019. PMID 35050996
- [Background] Beliveau M, Anderson D, Barker D, Kodihalli S, Simard E, Hall C, Richardson JS. Exposure-Response Modeling and Simulation to Support Human Dosing of Botulism Antitoxin Heptavalent Product. Clin Pharmacol Ther. 2022 Jul;112(1):171-180. doi: 10.1002/cpt.2620. Epub 2022 May 16. PMID 35467014
- [Background] Rao AK, Sobel J, Chatham-Stephens K, Luquez C. Clinical Guidelines for Diagnosis and Treatment of Botulism, 2021. MMWR Recomm Rep. 2021 May 7;70(2):1-30. doi: 10.15585/mmwr.rr7002a1. PMID 33956777